CLINICAL TRIAL: NCT03223662
Title: Metabolomic and BH3 Profiling of Esophageal Cancers: Identification of Novel Assessment Methods of Treatment Response for Precision Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left the NIH.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Caryn Steakley, R.N., Deputy Clinical Director, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170135; 17-C-0135
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Esophageal Cancer; Esophageal Adenocarcinoma; Esophageal Squamous Cell Cancer; Esophageal Neoplasms; Squamous Cell Carcinoma
Keywords: Neoadjuvant Chemoradiotherapy (nCRT); Esophagectomy; Tissue or serologic biomarkers
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Carcinoma, Squamous Cell | interventions — Chemoradiotherapy; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Chemoradiotherapy and esophagectomy (Other): Standard of care neoadjuvant chemoradiotherapy (nCRT) and esophagectomy
  Interventions: Other: Chemoradiotherapy; Procedure: Esophagectomy

INTERVENTIONS:
Other: Chemoradiotherapy — Chemotherapy: Carboplatin (AUC=2)x5 and Paclitaxel (50 mg/m(2))x5 for two cycles. Radiation: a total dose of 40.4 Gray (Gy) will be given in 23 fractions of 1.8 Gy, 5 fractions per week, starting the first day of the first cycle of chemotherapy.
Procedure: Esophagectomy — Minimally-invasive esophagectomy (RAMIE) or traditional open approach if necessary.

SUMMARY:
Background:

The number of patients with esophageal cancer keeps rising. For many patients, a combination of surgery, chemotherapy, and radiation is necessary to completely treat the disease. Usually, patients receive chemotherapy and radiation at the same time followed by surgery to remove the part of the esophagus with the tumor (Neoadjuvant chemoradiotherapy (nCRT)). Researchers want to learn how to make this treatment more effective.

Objective:

To see if biopsies before treatment can show which patients will do the best with a combination of chemotherapy, radiation, and surgery.

Eligibility:

Adults at least 18 years old with esophageal adenocarcinoma or squamous cell carcinoma who should be treated with chemotherapy, radiation, and surgery.

Design:

Patients will undergo standard testing that is routine for all patients with this disease. These tests include:

Medical history

Physical exam with activity and nutritional assessment

Standard lab tests

Imaging studies including a computerized axial tomography (CAT) scan and positron-emission tomography (PET) scan

Breathing test into a machine to measure size and function of lungs.

Biopsy for a small sample of tumor is removed by esophagogastroduodenoscopy (EGD): A tube inserted into the mouth under anesthesia

Endoscopic ultrasound is performed in some but not all patients.

Patients will have nCRT at the clinic or with their local doctor.

In 6 -12 weeks after nCRT, patients will undergo surgery with:

1. A robotically-assisted, minimally-invasive esophagectomy
2. Or, a traditional, open approach.

After surgery, patients are usually in the hospital for 2 weeks and have a feeding tube for at least 2 weeks and potentially longer until they are eating enough to not lose weight.

Patients will return for follow-up visits with labs and CAT scans every 6 months for the first two years then every year afterwards.

DETAILED DESCRIPTION:
Background:

* The incidence of esophageal cancer continues to increase with an estimated 16,900 new cases and 15,700 deaths in 2016. Esophageal adenocarcinoma (EAC) is the dominant histology in the United States and accounts for the rising incidence; the incidence of esophageal squamous cell cancer (ESCC) remains stable.
* Neoadjuvant chemoradiotherapy (nCRT) followed by esophagectomy is now a standard approach for locally advanced, operable esophageal cancer.
* A survival advantage compared to surgery alone was demonstrated in the phase III Chemo

Radiotherapy for Oesophageal cancer followed by Surgery Study (CROSS) trial.

* Patients who experience a pathological complete response (pCR) following neoadjuvant therapy are most likely to have long-term survival.
* Presently, accurate assessment of pathologic response requires esophagectomy. Positron-emissions tomography (fludeoxyglucose (FDG-PET)) and endoscopic evaluation with biopsies fail to detect cancer in a significant percentage of patients with residual disease following neoadjuvant therapy.
* Currently there are no validated tissue or serologic biomarkers which can be used to guide surgical management of esophageal cancer patients based on response to nCRT.

Primary Objective:

-To determine whether a metabolomic signature in tumor, blood, or urine or whether BH3 profiling of pre-neoadjuvant tumor biopsies correlates with the outcome of pathological complete response after neoadjuvant chemoradiotherapy for patients with esophageal adenocarcinoma or squamous cell carcinoma.

Eligibility:

-Patients with locally-advanced, histologically confirmed EAC or ESCC who are candidates for nCRT and esophagectomy.

Design:

* Patients will receive standard of care nCRT either at the National Cancer Institute (NCI) or at referring institutions.
* Specimens of plasma, urine, and esophageal tumor with matched normal esophagus will be obtained before neoadjuvant therapy for metabolomic profiling and BH3 profiling.

Blood, urine, normal esophagus, and tumor (if present) will be obtained after neoadjuvant therapy.

* Patients will undergo an esophagectomy as a robotically-assisted, minimally-invasive esophagectomy (RAMIE) or a traditional open approach for contraindications to minimally-invasive approaches or based on institutional expertise.
* Analysis will be performed to determine if pathological complete response (pCR) after chemoradiotherapy (CRT) correlates with pretreatment metabolomic signatures or BH3 profiling in tumor, blood or urine.
* Patients with EAC and ESCC will be evaluated independently.
* The accrual ceiling will be set to 120 patients for the entire study - 80 patients for EAC and 40 patients for ESCC to allow for unevaluable patients. The accrual is expected to be completed in 4 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed esophageal adenocarcinoma (EAC) or esophageal squamous cell carcinoma (ESCC).
* Disease should be deemed resectable by pre-operative computed tomography (CT) and/or positron-emission tomography (PET) scans and the patient should be operable based on surgeon assessment.
* Patients willing to complete neoadjuvant chemoradiotherapy (nCRT) per standard of care followed by esophagectomy. Patients will be treated under protocol 04-C0165.
* 18 years of age or older.
* Able to understand and sign the Informed Consent Document.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Patients must have organ and marrow function that is not prohibitive of surgical resection as defined below:

leukocytes greater than or equal to 3,000/mcL

absolute neutrophil count greater than or equal to 1,500/mcL

platelets greater than or equal to 50,000/mcL

* nCRT used in this study is potentially dangerous for developing human fetus. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration and 6 months post chemoradiotherapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Women must have a negative urine pregnancy test OR be post-menopausal for at least 2 years OR patient has had a hysterectomy

EXCLUSION CRITERIA:

* Patients in which nCRT followed by surgery is not the appropriate management:

  * Early stage disease that requires local therapy without chemoradiotherapy (CRT).
  * Patients with metastatic disease.
* Patients in which biopsy prior to starting nCRT is not obtainable.
* Patients who previously received neoadjuvant chemotherapy
* Concomitant medical problems in the opinion of physician that would place the patient at unacceptable risk for a major surgical procedure.
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, heart failure, hepatic disease that prohibits administration of neoadjuvant therapy or surgery.
* Women who are pregnant or breastfeeding because of the potentially dangerous effects of the chemotherapy on the fetus or infant.
* Patients with a diagnosis of another malignancy that is either active or in remission less than five years. Basal cell and squamous cell carcinoma of the skin are not contraindications to this protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Ripley, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piessen G, Messager M, Mirabel X, Briez N, Robb WB, Adenis A, Mariette C. Is there a role for surgery for patients with a complete clinical response after chemoradiation for esophageal cancer? An intention-to-treat case-control study. Ann Surg. 2013 Nov;258(5):793-9; discussion 799-800. doi: 10.1097/SLA.0000000000000228. PMID 24096755
- [Background] Stiles BM, Salzler G, Jorgensen A, Nasar A, Paul S, Lee PC, Port JL, Altorki NK. Complete metabolic response is not uniformly predictive of complete pathologic response after induction therapy for esophageal cancer. Ann Thorac Surg. 2013 Nov;96(5):1820-5. doi: 10.1016/j.athoracsur.2013.05.027. Epub 2013 Jul 26. PMID 23895888
- [Background] Shaikh T, Ruth K, Scott WJ, Burtness BA, Cohen SJ, Konski AA, Cooper HS, Astsaturov I, Meyer JE. Increased time from neoadjuvant chemoradiation to surgery is associated with higher pathologic complete response rates in esophageal cancer. Ann Thorac Surg. 2015 Jan;99(1):270-6. doi: 10.1016/j.athoracsur.2014.08.033. Epub 2014 Nov 18. PMID 25440267
- [Derived] Taylor Ripley R, Surman DR, Diggs LP, Trepel JB, Lee MJ, Ryan J, Davis JL, Steinberg SM, Hernandez JM, Hoang C, Kenney CM, Bond CD, Kunst TF, Letai A, Schrump DS. Metabolomic and BH3 profiling of esophageal cancers: novel assessment methods for precision therapy. BMC Gastroenterol. 2018 Jun 22;18(1):94. doi: 10.1186/s12876-018-0823-x. PMID 29933761

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Started | 2
Completed | 0
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Study closure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.55 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Metabolomic Signature in Tumor, Blood, or Urine and Outcome of Pathological Complete Response After Neoadjuvant Chemoradiotherapy in Patients With Esophageal Adenocarcinoma or Squamous Cell Carcinoma
Description: Specimens of normal esophagus, esophageal tumors, blood, or urine will be analyzed to determine specific signatures and outcome of pathological complete response after neoadjuvant chemoradiotherapy in patients with esophageal adenocarcinoma or squamous cell carcinoma. Response will be defined by the Mandard Score. Major response with no viable tumor (Grade 1) and <10% viable tumor (Grade 2) versus non major response of >10% viable tumor (Grade 3-5) as assessed by final pathology. Grade 1-2 is better survival than Grade 3-5.
Time Frame: After neoadjuvant therapy >4 weeks but prior to surgery
Population: Neither patient enrolled in the trial underwent resection based on post neoadjuvant therapy assessment of resectability. These patients were initially deemed potentially resectable prior to neoadjuvant therapy, but their course deviated from the initial plans. Therefore, the primary endpoint cannot be assessed.
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Number analyzed (Participants) | 0

2. Primary Outcome: BH3 Profiling of Pre-neoadjuvant Tumor Biopsy and Outcome of Pathological Complete Response After Neoadjuvant Chemoradiotherapy in Patients With Esophageal Adenocarcinoma or Squamous Cell Carcinoma
Description: Two tumor samples and two normal esophagus samples will be obtained for BH3 profiling of pre-neoadjuvant tumor biopsy and outcome of pathological complete response after neoadjuvant chemoradiotherapy in patients with esophageal adenocarcinoma or squamous cell carcinoma. Response will be defined by the Mandard Score. Major response with no viable tumor (Grade 1) and <10% viable tumor (Grade 2) versus non major response of >10% viable tumor (Grade 3-5) as assessed by final pathology. Grade 1-2 is better survival than Grade 3-5.
Time Frame: Pre-neoadjuvant therapy within 4 weeks, and after neoadjuvant therapy >4 weeks but prior to surgery
Population: as for outcome 1
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Number analyzed (Participants) | 0

3. Secondary Outcome: Metabolomic Profiles and B-cell Lymphoma (Bcl-2) Homology Domain-3 (BH-3) Profiling in Resectable Esophageal Adenocarcinomas (EAC) and Esophageal Squamous Cell Carcinoma (ESCC) Treated With Neoadjuvant Chemoradiotherapy (nCRT)
Description: Evaluation of metabolomic profiles and Bcl-2 homology domain-3 (BH-3) profiling in resectable esophageal adenocarcinomas (EAC) and esophageal squamous cell carcinoma (ESCC) treated with neoadjuvant chemoradiotherapy (nCRT)
Time Frame: Pre-neoadjuvant therapy within 4 weeks, and after neoadjuvant therapy >4 weeks but prior to surgery
Population: This outcome measure was not done. Neither patient enrolled in the trial underwent resection based on post neoadjuvant therapy assessment of resectability. These patients were initially deemed potentially resectable prior to neoadjuvant therapy, but their course deviated from the initial plans.
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Number analyzed (Participants) | 0

4. Secondary Outcome: Metabolomic Signatures or BH3 Profiling in Tumor, Blood, or Urine of Esophageal Adenocarcinoma (EAC) and Esophageal Squamous Cell Carcinoma (ESCC) With Major Responses (Mandard Score of 1 and 2) Versus Minimal Response (Mandard Score 3-5)
Description: Specimens of tumor, blood, or urine will be obtained to determine metabolomic signatures or BH3 profiling in tumor, blood, or urine of EAC and ESCC with major responses (Mandard score of 1 and 2) versus minimal response (Mandard score 3-5). Grade 1-2 is better survival than Grade 3-5.
Time Frame: Pre-neoadjuvant therapy within 4 weeks, and after neoadjuvant therapy >4 weeks but prior to surgery
Population: as for outcome 3
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Number analyzed (Participants) | 0

5. Secondary Outcome: Tumor Protein 53 (p53) Mutational Status and the Metabolomic Profiles
Description: One tumor sample and one normal esophagus sample will be obtained. p53 mutational analysis will be performed to determine mutational status and the metabolomic profiles .
Time Frame: Pre-neoadjuvant therapy within 4 weeks, and after neoadjuvant therapy >4 weeks but prior to surgery
Population: as for outcome 3
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Number analyzed (Participants) | 0

6. Secondary Outcome: Disease-free Survival in Esophageal Adenocarcinoma (EAC) and Esophageal Squamous Cell Carcinoma (ESCC) Patients Undergoing Neoadjuvant Chemoradiotherapy (nCRT) and Esophagectomy
Description: Disease-free survival is defined as the appearance of any new lesion that is likely metastatic or locally-recurrent esophageal cancer and will be assessed from the time of esophagectomy until development of metastatic disease or death, whichever comes first
Time Frame: From the time of esophagectomy until development of metastatic disease or death, whichever comes first
Population: This outcome measure was not done because one patient was deemed to be unsafe/unfit for surgery by the doctor. And the second patient was taken off-study prior to surgery because the principal investigator left the National Institutes of Health and closed the trial.
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival (OS) in Esophageal Adenocarcinoma (EAC) and Esophageal Squamous Cell Carcinoma (ESCC) Patients Undergoing Neoadjuvant Chemoradiotherapy (nCRT) and Esophagectomy
Description: Overall survival is defined as the time from treatment start date until date of death or date last known alive.
Time Frame: From treatment start date until date of death or date last known alive.
Population: as for outcome 6
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 23 days.
Description: There were no adverse events recorded for the participants on this trial during the time frame noted above.
Arm/Group | Neoadjuvant Chemoradiotherapy and Esophagectomy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT03223662/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT03223662/ICF_001.pdf